CLINICAL TRIAL: NCT03267719
Title: Intravaginal Laser Treatment of Mild and Moderate Stress Incontinence
Acronym: laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uro-Laser
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2019-03

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laser therapy (Experimental): Erbium-laser therapy will be applied
  Interventions: Device: laser therapy

INTERVENTIONS:
Device: laser therapy — Transvaginal erbium-laser treatment

SUMMARY:
The aim of the study is to evaluate the effectiveness of laser therapy as a non-surgical treatment option in patients with mild and moderate stress incontinence.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of laser therapy as a non-surgical treatment option in patients with mild and moderate stress incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Light or moderate stress incontinence
* mixed urine incontinence with predominance of the stress component
* written informed consent

Exclusion Criteria:

* Pregnancy
* patients treated radiotherapy in the small basin
* connective tissue disorders (e.g., Ehlers-Danlos syndrome, Marfan syndrome)
* patient with or after malignant disease of the uterus, ovaries, vagina and vulva
* former surgery due to stress incontinence (except for the patients who had a TVT insert with removal of the TVT)
* Descensus genitalis> POPQ Stage 1
* former surgery due to a genital lowering with vaginal netting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 month
  Quality of life will be access via ICIQ-SF questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Christl Reisenauer, Prof. Dr., Principal Investigator — University Women's Hospital Tübingen
Locations (1):
- Department for Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No